CLINICAL TRIAL: NCT06762665
Title: Impact of Interventional Radiology Consultation on the Spinal Infiltrations Effectiveness
Brief Title: RAdiology Consultation Effectiveness
Acronym: RACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL24_0113
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Radiology Interventional; Spinal Injections; Back Pain
Keywords: Consultation; Remote consultation; Radiology interventional; Spinal Injections; Health care
MeSH Terms: conditions — Back Pain | interventions — Injections, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Physical Consultation (PC) (Active Comparator): These patients have a consultation with the radiologist prior to the intervention, including an interview about their medical history and symptoms, a clinical examination, a review of the imaging file, an explanation of the procedure, and the opportunity to ask questions.
  Interventions: Procedure: Spinal injection; Other: pre-operative consultation
- Teleconsultation (TC) (Active Comparator): These patients have a teleconsultation with the radiologist prior to the intervention, including an interview about their medical history and symptoms, a review of the imaging file, an explanation of the procedure, and the opportunity to ask questions.
  Interventions: Procedure: Spinal injection; Other: pre-operative consultation
- No Consultation (NC) (Active Comparator): These patients not have a consultation prior to the procedure: The radiologist reviews the imaging file remotely. The explanation of the procedure is provided through documents, and questions are answered only on the day of the intervention.
  Interventions: Procedure: Spinal injection

INTERVENTIONS:
Procedure: Spinal injection — Patients underwent a spinal injection procedure under CT scan
Other: pre-operative consultation — Pre-operative consultation, in person or by teleconsultation, consists of an interview about the patient's history and symptoms. This is followed by a clinical examination and consultation of the patient's imaging file, to confirm the request for paraspinal infiltration and its location. In addition, the radiologist explains the procedure to the patient, supplementing the explanatory documents already provided at the time of the appointment, and outlines the results that may be expected and any complications.
  Arms: Physical Consultation (PC); Teleconsultation (TC)

SUMMARY:
Performing a consultation with the radiologist before a spinal invasive procedure serves to foster a trusting physician-patient relationship. It also provides an opportunity for the comprehensive explanation of the procedure, its aftermath, and any patient inquiries. We believe that this proactive approach has the potential to alleviate pre-procedure anxiety, thereby contributing to an enhanced overall experience of the intervention and its outcomes. Despite these potential benefits, it is noteworthy that such consultations are not systematically implemented, and their impact on the intervention effictness remains unexplored in existing literature.

The hypothesis is grounded in the belief that patients who perform a consultation preceding their spinal intervention are likely to witness improvements in both the overall experience of the procedure and its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Referred to the imaging department for a peri-spinal injection under CT guidance.
* Low back pain, dorsal pain, or neck pain with an average pain intensity of ≥ 5/10 on NPRS.

Exclusion Criteria:

* Patient unable to read and/or write French
* Patient unable to condut a teleconsultation (no phone, no internet connection)
* Current pregnancy, breastfeeding, or lack of effective contraception for women of childbearing age
* Lack of consent
* Legally protected population:

  * Adults protected by law (guardianship, curatorship, or judicial protection)
  * Non-emancipated minors
  * Individuals unable to express consent (research conducted in emergency situations)
  * Individuals deprived of liberty (by judicial or administrative decision, or involuntary hospitalization)
* Not affiliated with a social security scheme or not benefiting from such a scheme
* Participation in another research study with an ongoing exclusion period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the Numeric Pain Rating Scale (NPRS) between the 3 groups | 30 days after the surgical procedure
  Measuring pain on a numerical scale is a common method used to assess and communicate the intensity of a person's pain. The Numeric Pain Rating Scale (NPRS) is a numerical scale ranging from 0 to 10, where 0 represents no pain, and 10 represents the worst imaginable pain.
  Patients are asked to rate their pain by choosing a number that best reflects their current level of pain.
  Interpretation:
  0: No pain 1-3: Mild pain 4-6: Moderate pain 7-10: Severe pain

SECONDARY OUTCOMES:
Patient satisfaction with care | 30 days after the surgical procedure
  Satisfaction survey for healthcare is crucial to understanding the experiences of patients : The patient will be asked if he is satisfied:
  his medical care ( yes/no) If no : why and the arm to which he would have liked to belong
Assessment of Intervention Anxiety | Patient anxiety will be assessed at Day 0, just before the invervention
  The level of patient anxiety measured using a standardized anxiety scale (State-Trait Anxiety Inventory) The questionnaire includes 2 separate scales to assess state anxiety (how subjects feel now) and trait anxiety (how subjects usually feel). Each scale comprises 20 items.
  each item is rated from 0 to 3, so each scale is rated from 0 to 60, the higher the score, the greater the anxiety
Assessment of Medication Consumption | The Medication Consumption will be recorded throughout the study (120 days)
  The total quantity and frequency of analgesic, anti-inflammatory (NSAIDs), corticosteroid, and anxiolytic medications consumed by patients, recorded through patient self-reports and medical records.
Assessment of Procedure-Symptom Adequacy Improvement | before the procedure
  The percentage of procedures deemed fully adequate for the patient's symptoms and imaging, as determined by the radiologist's evaluation.
The Numeric Pain Rating Scale (NPRS) | To assess short-term pain 15 days after the surgical procedure
  Measuring pain on a numerical scale is a common method used to assess and communicate the intensity of a person's pain. The Numeric Pain Rating Scale (NPRS) is a numerical scale ranging from 0 to 10, where 0 represents no pain, and 10 represents the worst imaginable pain.
  Patients are asked to rate their pain by choosing a number that best reflects their current level of pain.
  Interpretation:
  0: No pain 1-3: Mild pain 4-6: Moderate pain 7-10: Severe pain
The Numeric Pain Rating Scale (NPRS) | To assess short-term pain 90 days after the surgical procedure
  Measuring pain on a numerical scale is a common method used to assess and communicate the intensity of a person's pain. The Numeric Pain Rating Scale (NPRS) is a numerical scale ranging from 0 to 10, where 0 represents no pain, and 10 represents the worst imaginable pain.
  Patients are asked to rate their pain by choosing a number that best reflects their current level of pain.
  Interpretation:
  0: No pain 1-3: Mild pain 4-6: Moderate pain 7-10: Severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Maxime PASTOR, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, Occitnaie, France

IPD SHARING:
Plan to Share IPD: Undecided